CLINICAL TRIAL: NCT05507710
Title: Indocyanine Green for Perfusion Assessment of DIEP Flaps: A Dutch Multicenter Randomized Controlled Trial
Brief Title: Indocyanine Green for Perfusion Assessment of DIEP Flaps
Acronym: FAFI
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, Alexander Vahrmeijer, Oncologic Surgeon - Hepatobiliary and Colorectal, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NL 68623.058.18
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Fat Necrosis
Keywords: Fat necrosis; Near-infrared fluorescence imaging; Indocyanine green; Free flap surgery; Breast reconstruction; Perfusion
MeSH Terms: conditions — Fat Necrosis

STUDY DESIGN:
Intervention Model Description: This is a two-armed randomized controlled trial:
  * interventional arm: evaluation of flap perfusion based on 1) clinical parameters, and 2) fluorescence imaging using ICG
  * conventional arm: evaluation of flap perfusion based on clinical parameters only
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant is blinded for the study arm. A second evaluator of postinterventional fat necrosis is blinded for the study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional study arm (Active Comparator): Surgery will be performed according to local protocol. Flap viability during adequate hemodynamic conditions is evaluated a standard of care. Then after anastomosis of the flap but before the inset, the second intervention is performed. Intervention: evaluation of the perfusion of the skin and fat with fluorescence imaging using ICG. The flap is marked according to the fluorescence imaging evaluation, and parts without perfusion are resected. The remaining flap is inset to the remaining breast skin.
  Interventions: Diagnostic Test: Near-infrared fluorescence imaging of perfusion
- Control arm (No Intervention): Surgery will be performed according to local protocol.Flap viability during adequate hemodynamic conditions is evaluated as standard of care. Then after anastomosis of the flap but before the inset, the surgeon will leave the room, the researcher will make a recording of the flap and this will have no consequences for the procedure.

INTERVENTIONS:
Diagnostic Test: Near-infrared fluorescence imaging of perfusion — Imaging with ICG near-infrared fluorescence is performed besides clinical judgement of the DIEP flap for perfusion evaluation. Based on fluorescence imaging, additional malperfused area(s) are resected.
  Arms: Interventional study arm

SUMMARY:
Currently during DIEP flap reconstruction, the perfusion of the flap is assessed by the clinical view of the surgeon. Identification of demarcated ischemic zones of the DIEP flap could be optimized by using fluorescence imaging with indocyanine green (ICG) in order to lower the rate of fat necrosis. This study evaluates whether intraoperative perfusion assessment with ICG fluorescence imaging causes a lower rate of fat necrosis compared to conventional intraoperative clinical evaluation of DIEP flaps.

DETAILED DESCRIPTION:
Rationale: Autologous breast reconstruction after mastectomy due to cancer or prophylactically due to genetically increased risk is frequently performed. A complication that may occur after a deep inferior epigastric artery (DIEP) reconstruction is the occurrence of fat necrosis in the transplanted flap due to ischemia (reperfusion injury). Identification of deep inferior epigastric artery perforators and identification of demarcated ischemic zones of the DIEP flap can be optimized by using fluorescence imaging with indocyanine green (ICG), as has been demonstrated in previous studies. This could result in less fat necrosis, less partial flap loss, and other complications. A randomized controlled trial would be the best study design to assess the value of ICG in determining the perfusion of DIEP flaps, thereby reducing the occurrence of fat necrosis and other complications.

Objective: To determine whether fluorescence imaging using ICG for the assessment of DIEP flap perfusion during surgery decreases the occurrence of fat necrosis compared to standard intraoperative clinical assessment of DIEP flap perfusion.

Study design: This is a two-armed randomized controlled trial:

* interventional arm: evaluation of flap perfusion based on 1) clinical parameters, and 2) fluorescence imaging using ICG
* conventional arm: evaluation of flap perfusion based on clinical parameters only

Study population: Patients scheduled for elective surgery for autologous breast reconstruction, uni- or bilateral, using DIEP or muscle sparing transverse rectus abdominis muscle (msTRAM) flaps. Female patients 18 years of age and older.

Intervention (if applicable): evaluation of flap perfusion based on 1) clinical parameters, and 2) fluorescence imaging using ICG

Main study parameters/endpoints: Difference in percentage of fat necrosis after autologous breast reconstruction using DIEP flaps between patients in whom fluorescence imaging was used and patients in whom flaps were clinically assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 years of age and older
2. Who underwent a mastectomy for breast cancer or prophylactic due to genetic predisposition
3. Patients scheduled for elective surgery for autologous breast reconstruction, uni- or bilateral, using DIEP or msTRAM flaps. In case of bilateral breast reconstruction the flaps should be bilateral anastomosed.
4. Written informed consent

Exclusion Criteria:

1. Allergy to ICG, iodine or shellfish
2. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the patient
3. Impaired renal function defined as eGFR< 50 mL/min/1.73m2 (this can be seen in the standard preoperative lab results)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical relevant fat necrosis | 3 months
  Clinically relevant fat necrosis is defined as a palpable mass, either painful or not, and with or without aesthetic complaints, and developed within three months after surgery. The following grading system according to Lie et al. is used. Only grade III till IV is classified as clinical relevant fat necrosis.
  III: Major compromised reconstructive outcome, flap involvement:15-50%, clinical findings: Major contour defects (multiple), surgical management: Debridement/secondary procedure IV: Subtotal poor reconstructive outcome, flap involvement: >50%, clinical findings: Skin defects, inadequate volume, volume loss, surgical management: Second local flap/ re-intervention initial flap

SECONDARY OUTCOMES:
Quantify perfusion of flaps | 3 months
  Based on NIRF recordings and correlate these to the development of fat necrosis.
Registration of re-interventions | 3 months
  necessary to treat fat necrosis, in numbers and percentages
Registration of postoperative complications | 3 months
  in numbers and percentages
Duration of surgery in minutes | 1 day
  Of all surgical procedures included
Percentage extra resected tissue | 1 day
  of initial flap in grams based on perfusion assessment
Personal experience/opinion of surgeon performing surgery with fluorescent imaging using ICG. | 1 day
  After every surgery the NASA TASK Load Index is taken by the surgeon.
Patient satisfaction | 3 months
  using BREAST-Q questionnaire, this is an validated questionnaire that is used in multiple research for measuring patient satisfaction

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Erasmus Medical Center, Rotterdam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tange FP, Verduijn PS, Sibinga Mulder BG, van Capelle L, Koning S, Driessen C, Mureau MAM, Vahrmeijer AL, van der Vorst JR. Near-infrared fluorescence angiography with indocyanine green for perfusion assessment of DIEP and msTRAM flaps: A Dutch multicenter randomized controlled trial. Contemp Clin Trials Commun. 2023 Apr 2;33:101128. doi: 10.1016/j.conctc.2023.101128. eCollection 2023 Jun. PMID 37091505